CLINICAL TRIAL: NCT01298115
Title: Patient Information About Options for Treatment of Stage 5 Chronic Kidney Disease
Brief Title: Patient INformation About Options for Treatment - PINOT
Acronym: PINOT
Status: Completed | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); Sydney South West Area Health Service (Other Government); South West Sydney Local Health District (Other)
Responsible Party: A/Prof Kirsten Howard, University of Sydney
Other Study IDs: RM-1/09
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease; dialysis; pre dialysis education; transplantation; conservative care
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stage 5 chronic kidney disease: Incident patients commencing renal replacement therapy or conservative care

SUMMARY:
This prospective observational study is designed to find out what treatment options new patients with chronic kidney disease learn about from their renal unit.

Aims: To determine the proportion of new CKD patients who receive information about treatment options prior to commencing dialysis, pre-emptive transplantation or conservative management. To determine the timing (i.e. patient's stage of disease) when information is given. To find out whether patients have a friend or family member with them when information is given.

Research Design and methods: This study is an assessment of CKD education practices. Nephrologists and pre-dialysis coordinators from each renal unit will complete questionnaires about information that was given to each new dialysis, pre-emptive transplant or conservatively managed patient that started treatment during a 3 month period.

Study hypothesis: Approximately one third of CKD patients will receive information after starting treatment. There will be a positive association between in-centre haemodialysis and later referral, non-English speaking background, and advancing age. Significance: The results from this national audit will provide Australian nephrologists and renal nurses with evidence about CKD education practices and compliance with clinical practice guidelines. The results may highlight opportunities for improvement in practice.

DETAILED DESCRIPTION:
Additional research objectives and key research questions:

1. To determine the proportion of patients who receive information about: pre-emptive transplantation; peritoneal dialysis; home haemodialysis; centre based haemodialysis; supported non-dialytic care or conservative management.

3. To determine the proportion of incident patients that have a non-English speaking background (NESB) requiring an interpreter or translated materials.

4. To examine associations between age, gender, health insurance status, NESB, CKD stage and information provided on initial treatment commenced.

5. To determine the proportion of patients who choose not to dialyse.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Australian adult or pediatric renal units
* Patients with Stage 5 chronic kidney disease commencing dialysis or having a pre-emptive transplant or with decision made for conservative care and eGFR < 15ml/min/1.73m2 between 1st July and 30th September 2009

Exclusion Criteria:

* Patients with acute kidney injury not requiring chronic renal replacement therapy
* Patients with a failing kidney transplant returning to dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with chronic kidney disease attending renal treatment centres in Australian public hospitals and private practices.
Sampling Method: Probability Sample
Enrollment: 721 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of incident Stage 5 CKD patients who receive information about their treatment options prior to commencing treatment | Time prior to commencement of treatment. eg. 3 months

SECONDARY OUTCOMES:
Stage of CKD (based on eGFR) when information about treatment options is first given | one time point prior to commencement of treatment
Patient and unit characteristics associated with commencing renal replacement therapy versus conservative care | One time point based on commencement date of first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Howard, PhD, Study Chair — University of Sydney
Locations (1):
- University of Sydney, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Morton RL, Howard K, Webster AC, Snelling P. Patient information about options for treatment: Methods of a national audit of information provision in chronic kidney disease. Nephrology (Carlton). 2010 Sep;15(6):649-52. doi: 10.1111/j.1440-1797.2010.01340.x. PMID 20931747
- [Result] Morton RL, Howard K, Webster AC, Snelling P. Patient INformation about Options for Treatment (PINOT): a prospective national study of information given to incident CKD Stage 5 patients. Nephrol Dial Transplant. 2011 Apr;26(4):1266-74. doi: 10.1093/ndt/gfq555. Epub 2010 Sep 6. PMID 20819955